CLINICAL TRIAL: NCT05854303
Title: Prospective Evaluation of the Effect of Opioid Cessation on Opioid-Induced Esophageal Dysfunction (OIED)
Brief Title: Effect of Opioid Cessation on Opioid-Induced Esophageal Dysfunction
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Diana L. Snyder, Principal Investigator, Mayo Clinic
Other Study IDs: 23-001879
Record Dates: First submitted 2023-05-03; First posted 2023-05-11 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: Opioid-Induced Esophageal Dysfunction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Opioid Cessation: Subjects able to complete opioid cessation.
  Interventions: Behavioral: Opioid cessation
- Non-Opioid Cessation: Subjects unable to complete opioid cessation.
  Interventions: Other: No opioid cessation

INTERVENTIONS:
Behavioral: Opioid cessation — opioid cessation will occur during pain rehabilitative program over approximately 3 weeks
  Groups: Opioid Cessation
Other: No opioid cessation — Subjects will not stop taking opioids
  Groups: Non-Opioid Cessation

SUMMARY:
The purpose of this study is to evaluate the effect of opioid cessation on opioid-induced esophageal dysfunction (OIED).

ELIGIBILITY:
Inclusion Criteria:

- Patients enrolled in the Pain Rehabilitation Center for opioid cessation, with or without esophageal symptoms.

Exclusion Criteria:

* Inability to provide informed consent.
* Patients with previous gastroesophageal surgery or pneumatic dilation.
* Esophageal botulinum toxin injection within the prior 12 months.
* Esophageal stricture
* Achalasia types I and II
* Allergy to Lidocaine or other local anesthetics
* Subjects on anticoagulation
* Bilateral nasal obstruction
* Pregnancy or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients being seen in the Pain Rehabilitation Center for opioid cessation at Mayo Clinic Rochester.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Estimated)
Dates: Start 2023-09-18 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Number of subjects to have opioid-induced esophageal dysfunction resolution | 4 weeks
  Number of subjects to have resolution of opioid-induced esophageal dysfunction

SECONDARY OUTCOMES:
Number of subjects with dysphagia | 4 weeks
  Number of subjects that are chronic opioid users presenting to an opioid cessation clinic to have dysphagia
Number of subjects with chest pain | 4 weeks
  Number of subjects that are chronic opioid users presenting to an opioid cessation clinic to have chest pain
Number of subjects with opioid-induced esophageal dysfunction | 4 weeks
  Number of subjects that are chronic opioid users presenting to an opioid cessation clinic to have opioid-induced esophageal dysfunction

CONTACTS AND LOCATIONS:
Overall Officials: Diana Snyder, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Minnesota, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials